CLINICAL TRIAL: NCT01700088
Title: The Effect of Nasal Cannulae During the First 2 Hours Postoperative in Patient
Brief Title: The Effect of Nasal Cannulae During the First 2 Hours Postoperative in Patient Undergoing Thoracotomy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Other Study IDs: 541/2555(EC2)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Hypoxia; Post Pulmonary Resection
Keywords: hypoxemia; Post Pulmonary Resection
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oxygen cannular: After lung resection surgery,every patient will received supplementary oxygen 5 L/minutes via oxygen cannular for 120 minutes

SUMMARY:
At our institute,during the first 2 hour postoperative, we used to give supplement oxygen via face mask in patient having lung resection surgery. After then if the patient is fine, we'll replace the face mask with nasal cannular untie the next morning. We hypothesized that oxygen mask can be replace by nasal cannular without any hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 18 years old
* Patient undergoing lobectomy or pneumonectomy or wedge resection
* ASA 1-3
* Preoperative oxygen saturation < 95 %

Exclusion Criteria:

* Cannot communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing lung resection surgery.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 30 minutes
  We continuously monitor oxygen saturation and record every 5 minutes for 30 minutes postoperative.

SECONDARY OUTCOMES:
Incidence of hypoxemia | 3 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand